CLINICAL TRIAL: NCT01931943
Title: A Phase Ib Study to Evaluate the Tolerability and Pharmacokinetics of Selatinib Ditosilate Tablets in Patients With Advanced Breast Cancer
Brief Title: A Phase Ib Study of Selatinib Ditosilate Tablets in Patients With Advanced Breast Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QLSLTN-102
Record Dates: First submitted 2013-08-25; First posted 2013-08-30 (Estimated); Last update posted 2013-08-30 (Estimated); Status verified 2013-08

CONDITIONS: Advanced Breast Cancer

ARMS (1):
- Selatinib Ditosilate Tablets (Experimental): Selatinib Ditosilate either at 450,750,1000,1250mg, p.o. once daily
  Interventions: Drug: selatinib ditosilate tablets

INTERVENTIONS:
Drug: selatinib ditosilate tablets

SUMMARY:
Brief Description:

This study is designed to evaluate the safety and tolerability of oral Selatinib Ditosilate Tablets, and explore the maximum tolerated dose (MTD) and dose-limiting toxicity in patients with advanced breast cancer.

DETAILED DESCRIPTION:
1. To evaluate the safety and tolerability of oral Selatinib Ditosilate Tablets, and explore the maximum tolerated dose (MTD) and dose-limiting toxicity (DLT).
2. To determine the pharmacokinetic profile of single and multi oral Selatinib Ditosilate Tablets .
3. To determine preliminary dose and regimen for phase II study of oral Selatinib Ditosilate Tablets.
4. To assess preliminary antitumor activity .

ELIGIBILITY:
Inclusion Criteria:

* women aged 18-65.
* Patients with ECOG performance status of 0 or 1.
* Expected life-expectancy of more than 3 months.
* Patients must have histologically or cytologically confirmed breast cancer. Either the primary breast tumor or the metastasis must overexpress HER2; acceptable methods of measurement of HER2 expression include immunohistochemistry (IHC) and fluorescence in situ hybridization (FISH); tumors tested by IHC must be 3+ positive for HER2 overexpression immunohistochemistry ; tumors tested by FISH must be positive.
* Prior Herceptin therapy is discontinued because of disease progression or patients can not afford for Herceptin therapy.
* patients with at least one measurable lesion (RECIST1.1 criteria).
* Hematology： WBC≥3.5×109/L, ANC≥1.5×109/L, PLT≥100×109/L，HB≥90g/L;
* Biochemistry： Serum bilirubin≤1.5 times upper limit of normal (ULN),AST and ALT ≤1.5 times ULN; creatinine and urea nitrogen≤1.5 times ULN; LVEF≥50%, ECG normal, and Fridericia corrected QT(QTcF)<470ms.
* patients receiving damage caused by other therapeutic has been restored, the interval more than six weeks since the last receiving nitroso or mitomycin; more than 4 weeks since last receiving radiotherapy, other cytotoxic drugs or surgery.
* Subjects can swallow and have normal gastrointestinal function.
* Female subjects should agree to take contraceptives during the study and within 6 months after the study (such as intrauterine device [IUD], contraceptive drugs or condoms); within 7 days before they enter the study, their serum or human chorionic gonadotropin should be negative, and must be in the non-lactation period.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients have uncontrolled large pleural effusion and ascites.
* Patients have received steroid for more than 50 days, or requiring for steroid therapy for a long time.
* Requirement for the therapeutic drugs prolonging QT interval(such as anti-arrhythmia drugs), and can not interrupt them.
* Patients with a history of symptomatic brain metastases.
* Patients have received small molecule targeted drug therapy of inhibition of HER-2 or EGFR.
* Patients have participated in other drug clinical research in the past 4 weeks.
* Pregnant or lactating women are excluded from this study.
* Patients with a history of allergic reactions attributed to compounds of similar chemical composition to the agents used in the study are ineligible;
* Patients with active infection ;
* Patients with cardiac disease including Angina, any significant or need to be treated arrhythmia，Myocardial infarction, Heart failure, LVEF<45%, other heart diseases that are not suitable for participating in the study judged by investigator.
* Patients with other concurrent severe and/or uncontrolled medical conditions （including hypertension, severe diabetes, thyroid disease, etc.) that could cause unacceptable safety risks or compromise compliance with study requirements are ineligible.
* Patients with a history of mental disorders, including epilepsy or dementia are ineligible.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2013-04; Primary Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity(DLT) | 21 days
Maximum tolerated dose(MTD) | 21 days

SECONDARY OUTCOMES:
Pharmacokinetics | 21 days
  Selatinib Ditosilate pharmacokinetic parameters , include AUC, Cmax, Tmax, and t1/2
Pharmacodynamics | 7 weeks
  The response of Salatinib Ditosilate on tumor measured by CT or MRI.

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Institute and Hospital,Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Zhang T, Li Q, Chen S, Luo Y, Fan Y, Xu B. Phase I study of QLNC120, a novel EGFR and HER2 kinase inhibitor, in pre-treated patients with HER2-overexpressing advanced breast cancer. Oncotarget. 2017 May 30;8(22):36750-36760. doi: 10.18632/oncotarget.13581. PMID 27902470